CLINICAL TRIAL: NCT04662034
Title: Prospective, Randomized, Open, Comparison Study to Demonstrate the Performance and the Safety of Cardiac Microcurrent Therapy (C-MIC) System
Brief Title: Performance and Safety of the Cardiac Microcurrent Therapy System
Acronym: C-MIC-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berlin Heals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMIC-II
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-03

CONDITIONS: Systolic Left Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Standard of Care

STUDY DESIGN:
Masking Description: Device vs Standard of Care, no masking possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Device plus Standard of Care (Experimental): Device plus Standard of Care
  Interventions: Device: CMIC; Drug: Standard of Care (SOC)
- Standard of Care (Other): Standard of care drug treatment
  Interventions: Drug: Standard of Care (SOC)

INTERVENTIONS:
Device: CMIC — The C-MIC System consists of three implantable parts: a transvenous and an epicardial lead which are both connected to an implanted power source, and an external programing device. The patch lead is placed over the free wall of the left ventricle and fixated with sutures. When lead placement is achieved, the leads are then tunneled subcutaneously to the infraclavicular region and connected to the power source.
  Arms: Device plus Standard of Care
Drug: Standard of Care (SOC) — Patients receive optimal SOC based defined in pertinent guideline and at the discretion of the investigator
  Other Names: Standard drug therapy

SUMMARY:
Patients with idiopathic dilative cardiomyopathy who have systolic left ventricular dysfunction (NYHA III - IV) despite adequate therapy according to treatment guidelines of heart failure and who have a baseline left ventricular ejection fraction of ≥25% and ≤35 will receive a C-MIC System and microcurrent therapy after device implantation with optimal medical management. At the end of the study after 6 months, the C-MIC System will be turned off. The control group will receive optimal medical management without device implantation.

DETAILED DESCRIPTION:
Target patients for the C-MIC System are patients with idiopathic dilative cardiomyopathy who have systolic left ventricular dysfunction (NYHA class III - NYHA class IV) despite adequate therapy of heart failure and a left ventricular ejection fraction ranging from 25% to 35% with a history of heart failure of more than 1 year but less than 5 years.

The study's objective is to determine the safety and effectiveness of C-MIC therapy in patients with moderate to severe heart failure under optimal medical therapy. Data from a pilot study (C-MIC-I) indicate that an increase of ≥ 8% of the left ventricular ejection fraction can be achieved within a treatment period of 6 month. Therefore, the study hypothesis assumes hat the change in LVEF from baseline to 6 months will be significantly greater in patients undergoing C-MIC therapy (device group) in addition to guideline directed medical therapy (GDMT) compared patients remaining on GDMT alone (control group).

Subjects will be randomized in a 1:1 ratio to receive the C-MIC System in addition to optimal medical management or to receive optimal medical management alone without device. Due to the risks associated with the implantation, a sham (placebo) procedure is not warranted.

The primary endpoint will be measured as the difference in the change in LVEF from baseline to 6 months, measured via cardiac ultrasound and expressed in percentage. LVEF measurements will be compared between the device and control groups and verified by a core lab at baseline, week 4, month 4 and month 6.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic dilative cardiomyopathy who have systolic left ventricular dysfunction despite of adequate therapy of heart failure (NYHA III - IV (ambulatory)).
* Patients with symptomatic chronic heart failure for more than 1 year and less than 5 years at screening.
* Patients who have a baseline left ventricular ejection fraction of ≥25% and ≤35% assessed by echocardiography within 30 days prior to study inclusion.
* Patient who understands the nature of the procedure and on-going device therapy. Patient is informed about their participation in a chronic human study and about the intended treatment period of 6 months which is derived by the fact that according to current knowledge microcurrent treatment exceeding 6 months will not have additional favorable effects which means will not further improve cardiac function. Accordingly, battery life is limited. Furthermore, the patient is informed about the possibility for device explantation, informed regarding possible risks and is able to give written informed consent prior to any procedures and is considered willing and able to adhere to study regimen and to return for all follow-up visits.
* Patients are receiving guideline conform heart failure therapy
* Patients receiving appropriate, stable guideline conform anti-heart failure therapy during the 3 months prior study inclusion (OMM). Stable is defined as no more than a 50% increase or 50% decrease in dose. If the patient is intolerant to full anti-heart failure medication, documented evidence must be available.
* Patients who are able to perform a 6-minute walk test.
* Patients must have a body mass index within the range of 20 - 36 kg/m².
* Informed consent in writing from patient.
* Patients with an ICD systems can be included providing patients are not pacemaker dependent and the ICD system uses a single coil electrode the leads can be implanted in such a way that it is ensured, that the metal parts of the coil electrodes do not touch each other.

Exclusion Criteria:

* Patients who have a potentially correctible cause of heart failure, such as valvular heart disease or congenital heart disease.
* Patients with an indication for a CRT system according to current guidelines.
* Patients who have been hospitalized for heart failure which required the use of inotropic support within 30 days before enrollment.
* Patients with systolic blood pressure above 150 mmHg and diastolic blood pressure above 90 mmHg despite optimal antihypertensive medical treatment.
* Patients with hemoglobin blood level < 12 g/dl in male and < 10 g/dl in female patients.
* Patients with primary pulmonary hypertension
* Patients who have a genetic connective tissue disease (for example Marfan syndrome).
* Patients with constrictive pericarditis.
* Patients with a prosthetic tricuspid valve.
* Patients in whom access for implantation of the leads cannot be obtained (i.e., known venous occlusion, post radiation therapy).
* Patients who have other preexisting epicardial leads.
* Patients who have undergone prior heart surgery.
* Patient with other features (i.e., thorax deformity) that in the eyes of the investigator make the straightforward placement of the device seem unlikely.
* Patients with an ICD system who are pacemaker dependent
* Patients with an ICD system with a dual coil electrode.
* Patients with a CRT system or pacemaker.
* Patients with a CCM system.
* Current pregnancy or
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception (e.g., intrauterine device, oral contraceptives, barrier methods, or other contraception deemed adequate by the investigator) 2 months before and until 1 month after C-MIC therapy.
* Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 2 months before screening.
* Breastfeeding/lactating women
* Patients whose exercise tolerance is limited by a condition other than heart failure (e.g., chronic obstructive pulmonary disease, peripheral vascular disease, orthopedic or rheumatologic conditions) or who are unable to participate in a 6-minute walk test.
* Patients on immunosuppressive therapy.
* Patients with present malignancy.
* Patients with an active infection considered by the investigator to be unsafe for the patient's participating in the trial.
* Patients with renal dysfunction (i.e., estimated glomerular filtration rate <45 mL/min / 1,73 m²)
* Patients with history or presence of relevant liver diseases or hepatic dysfunction as indicated by abnormal liver function tests at screening and baseline: ALT (SGPT), AST (SGOT), γ-GT, alkaline, phosphatase and serum bilirubin > 2 × upper limit of normal (ULN). Increase of these liver enzymes caused by cardiac disorders in the absence of other possible causes of liver damage are not are not meant by this.
* Patients with a history of drug or alcohol abuse within the 12 months prior to screening.
* Patients who, in the opinion of the Principal Investigator, are unlikely to comply with the protocol requirements, instructions and trial related restrictions, e.g., uncooperative attitude, inability to return for follow-up visits, psychological illness, and improbability of completing the trial.
* Participation in any study of an investigational device or drug within 90 days prior to planned study.
* Vulnerable Patients (e.g., patients requiring a legal representative, patients kept in detention, any service within the army, and employees of the sponsor or at an investigator site).
* Patients who are not able to avoid the following areas (i.e., due to work) such as areas with strong magnetic fields, areas with strong external electrical influences, areas with a warning notice "Access prohibited for pacemaker patients" or similar and areas with high temperatures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Performance | 6 months
  Change of the left ventricular ejection fraction (LVEF) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Peter Goettel, MD, Study Director — Berlin Heals GmbH
Locations (20):
- Bosnia and Herzegovina (2):
  - University Clinic, Banja Luka
  - University Clinic Sarajevo, Sarajevo
- Diagnostic and Consultative Center Neoclinic Ead, Sofia, Bulgaria
- Clinical Hospital Dubrava, Zagreb, Croatia
- HNA Homolce Hospital, Prague, Czech Republic, Czechia
- Germany (5):
  - German Heart Center Charité, Berlin
  - Vivantes Humbold Clinic, Berlin
  - Heart Center Dresden, Dresden
  - Medical University Hannover, Hanover
  - University Hospital Regensburg, Regensburg
- St. Luke´s Hospital, Thessaloniki, Greece
- University Clinic Skopje, Skopje, North Macedonia
- Poland (2):
  - Polish-American Heart Clinic, Bielsko-Biala
  - University Hospital Wroclaw, Wroclaw
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Institute of Cardiovascular Diseases Dedinje, Belgrade
  - Institute of Cardiovascular Diseases, Kamenitz
- Bellvitge University Hospital, Barcelona, Spain
- Universitaetsspital Basel, Basel, Switzerland

REFERENCES:
- [Result] Rame JE, Schmitto JD, Kosevic DN, Kovacevic-Preradovic T, Jovev S, Zdravkovic M, Granov N, Popov T, Rudez I, Vukovic P, Ristic V, Neuzil P, Holtdirk A, Ruhparwar A, Khan MS, Dungen HD, Brandes K, Goettel P, Mueller J, Kallel F, Friede T, Peric M, Fudim M, Anker SD; C-MIC II Trial Investigators. Cardio-microcurrent device treatment for heart failure with reduced ejection fraction: Results from the C-MIC II open-label randomized controlled trial. Eur J Heart Fail. 2025 Oct;27(10):1837-1849. doi: 10.1002/ejhf.3763. Epub 2025 Jul 15. PMID 40660878